CLINICAL TRIAL: NCT01910012
Title: Phase 2 Study of ADI-PEG 20 in Acute Myeloid Leukemia
Brief Title: PH 2 ADI-PEG 20 Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Polaris Group (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POLARIS2012-001
Record Dates: First submitted 2013-07-10; First posted 2013-07-29 (Estimated); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Acute Myeloid Leukemia
Keywords: Argininosuccinate Synthetase; Arginine; Arginine deiminase; Failed prior systemic therapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — ADI PEG20; Polyethylene Glycols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ADI-PEG 20 (Experimental): arginine deiminase formulated with polyethlene glycol
  Interventions: Drug: ADI-PEG 20

INTERVENTIONS:
Drug: ADI-PEG 20
  Other Names: arginine deiminase formulated with polyethylene glycol

SUMMARY:
Certain cancers require the amino acid arginine. Arginine deiminase (ADI) is an enzyme from microbes that degrade arginine. ADI has been formulated with polyethylene glycol and has been used to treat patients that have cancers that require arginine. In this study, the investigators will evaluate the response rate, as determined by the revised International Working Group recommendations.

ELIGIBILITY:
Inclusion Criteria:

1. Acute myeloid leukemia (AML) diagnosed by morphologic, histochemical or cell surface marker criteria.
2. Patients with AML must have either:

   (a) relapsed or refractory leukemia after receiving at least one prior conventional induction therapy. Those in early first relapse must not have a matched donor and/or they must not be a candidate for allogeneic stem cell transplantation (usually this would mean the patient is too ill, obese, has a co-morbid condition or is over the age of 55 years) or (b) poor-risk AML as defined below: (i) Treatment related AML, except if it is associated with favorable cytogenetics (e.g., inversion 16, t(16;16), t(8;21), t(15;17), and not a candidate for stem cell transplantation, or (ii) AML with an antecedent hematologic disease (e.g., MDS, myelofibrosis, polycythemia vera, etc.), and not a candidate for stem cell transplantation.

   (iii) De novo AML > 70 years of age. (iv) AML with unfavorable cytogenetics regardless of age (>18 years), if patients are not candidates for allogeneic transplantation. Unfavorable cytogenetics are the following: complex (>3 abnormalities), -7, -5, 7q-, 5q-, abnormalities of 11q23 excluding t(9;11), t(9;22), inversion 3, t(3;3), t(6;9).

   (c) Patients older than 60 years of age who had AML (i.e., > 20% bone marrow blasts) and no prior therapy for AML
3. Age ≥ 18 years.
4. ECOG performance status of 0-2.
5. Post-menarche female subjects and male subjects must be asked to use appropriate contraception for both the male and female for the duration of the study. Subjects must agree to use two forms of contraception or agree to refrain from intercourse for the duration of the study. Females must not be pregnant at the start of the study, and a serum human chorionic gonadotropin (HCG) pregnancy test must be negative before entry into the study.

Exclusion Criteria:

1. Patients with infections requiring intravenous (IV) antibiotic/antiviral therapy are not eligible for entry onto the study; patients on prophylactic antibiotics or antivirals are acceptable.
2. Pregnancy or lactation.
3. Expected non-compliance.
4. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure (New York Heart Association Class III or IV), cardiac arrhythmia, psychiatric illness, social situations that would limit compliance with study requirements or DIC.
5. Subjects who have had any anticancer treatment prior to entering the study and have not recovered to baseline (except alopecia) or≤ Grade 1 AEs, or deemed irreversible from the effects of prior cancer therapy. AEs > Grade 1 that are not considered a safety risk by the Sponsor and investigator may be allowed upon agreement with both.
6. Subjects with history of another primary cancer, including co-existent second malignancy, with the exception of: a) curatively resected non-melanoma skin cancer; b) curatively treated cervical carcinoma in situ; or c) other primary solid tumor with no known active disease present in the opinion of the investigator will not affect patient outcome in the setting of current diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2015-01-06 (Actual); Primary Completion 2016-09-12 (Actual); Study Completion 2017-05-05 (Actual)

PRIMARY OUTCOMES:
Response Rate | 2 years estimated

SECONDARY OUTCOMES:
Safety and tolerability | 2 years estimated
  * Time on treatment
  * Overall survival
  * Evaluate the response rate and correlate with patient disease burden, and type of disease.
  * Determine the pharmacodynamics of ADI-PEG 20
  * Determine the immunogenicity of ADI-PEG 20

CONTACTS AND LOCATIONS:
Locations (6):
- MD Anderson, Houston, Texas, United States
- Taiwan (5):
  - Chang Gung Medical Foundation-Kaohsiung, Kaohsiung City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - CMUH, Taichung
  - NCKUH, Tainan
  - CGMH-LK, Taoyuan District

REFERENCES:
- [Derived] Tsai HJ, Jiang SS, Hung WC, Borthakur G, Lin SF, Pemmaraju N, Jabbour E, Bomalaski JS, Chen YP, Hsiao HH, Wang MC, Kuo CY, Chang H, Yeh SP, Cortes J, Chen LT, Chen TY. A Phase II Study of Arginine Deiminase (ADI-PEG20) in Relapsed/Refractory or Poor-Risk Acute Myeloid Leukemia Patients. Sci Rep. 2017 Sep 12;7(1):11253. doi: 10.1038/s41598-017-10542-4. PMID 28900115